CLINICAL TRIAL: NCT04739332
Title: Assessing the Effect of the Newborn Behavioral Observations System on Maternal Sensitivity Four Months Post-partum
Brief Title: The Effect of the Newborn Behavioral Observations System on Maternal Sensitivity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Center for Parents and Infants, Iceland (Other)
Collaborators: The Icelandic Nurses' Association (Unknown); Health care of the capital area, Iceland (Unknown); Research and Analysis, v/University of Reykjavik (Unknown); Regionsenter for barn og unges psykiske helse, Norway (Unknown)
Responsible Party: Principal Investigator, Stefania Birna Arnardottir, Family nurse specialist, MSc, Center for Parents and Infants, Iceland
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CParentsInfants
Record Dates: First submitted 2020-12-17; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Mother-Infant Interaction
Keywords: perinatal depression; maternal sensitivity; Infant emotion regulation

STUDY DESIGN:
Intervention Model Description: RCT
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NBO intervention for at-risk mothers (Experimental): NBO intervention for at- risk mothers. 3 NBO sessions added to the routine follow-up delivered once per week during the first month postpartum. The intervention is delivered by a nurse certified in the NBO system.
  Interventions: Behavioral: The Newborn behavioral observations system
- Treatment as usual (No Intervention): Participants receive 3 routine follow-up by the local health visitor/midwife during the first month

INTERVENTIONS:
Behavioral: The Newborn behavioral observations system — The NBO system is a relationship building tool to enhance parental sensitivity in the newborn period. Mothers at risk for post-partum depression are supported by a clinician to respond with confidence to their newborn's individual needs.
  Arms: NBO intervention for at-risk mothers

SUMMARY:
The study evaluates if the Newborn Behavioral Observation system, a relationship building tool, delivered to at risk mothers will have, on one site, an effect on maternal sensitivity and the other site on Childs responsiveness, measured by the Emotional Availability (EA) Scales at 4 months post partum.

DETAILED DESCRIPTION:
The aim of this study is to evaluate the effect of the Newborn Behavioral Observation (NBO) on one site, on maternal sensitivity and on other site on Childs responsiveness, assessed by EAS at 4 months post partum. The NBO intervention serves to sensitize parents to the infant's capacities and individuality and to enhance the parent-infant relationship by strengthening parents 'confidence and practical skills in caring for their infants.

The study will use a RCT design. The NBO intervention group will be compared with a control group who will receive usual post partum care offered by primary health care in Reykjavik, Iceland. Inclusion criteria are pregnant women with an EPDS sum score above 9 in the third trimester and/or a previous history of trauma, anxiety and depression.

The NBO intervention group (n=30) will receive three home visits during the 2nd to 4th week after birth in addition to their usual home visits. The control group (n=30) will receive regular follow-up (without NBO sessions). At 4 months all participating mothers will be videotaped during daily caring, feeding or play episodes with their infant.

Baseline questionnaire (T1) contained information on household income, parity, education level and the number of children living in the household. Maternal depressive symptoms were measured by the Icelandic version of The Edinburgh Postnatal Depression Scale (EPDS) at 24-28 weeks of gestation (T0), six weeks postpartum (T5) and again at 4 months postpartum (T6). The EPDS is a 10-item self-report scale that assesses current (last week) postpartum depressive symptomatology. Each item is rated on a 4-point scale (0-3), yielding a total score ranging from 0 to 30, with higher scores indicating increased symptomatology of postpartum depression.

The videos will be coded by use of the The Emotional Availability (EA) Scale to assess maternal sensitivity and Childs responsiveness. The EA Scale consists of six dimensions of emotional availability in the relationship: four for the adult (sensitivity, structuring, nonintrusiveness and nonhostility) and two for the child (responsiveness to adult and involvement of adult). The EA direct score for the first dimension, sensitivity for mothers and responsiveness for the child, is reported. The score seven (range 1-7) is the highest/best possible score on the two first catagories and three (range 1-3) is the higest/best score fot the next five catargories. This seven catagories in each domain make the direct score, witch can reach from 7-29 where the 29 is the higest. In addition to the 6 diementions the Clinical Screeners....... The EA Scale is validated in various settings and cultures and will serve as the main outcome measure in the RCT.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women and their partners
* Age of 18 or more.
* Understanding Icelandic.
* Having score of EPDS scale of more than 9 or history of depression and/or anxiety

Exclusion Criteria:

* Not speaking or understanding Icelandic.
* Having given birth within 35 weeks of pregnancy.
* Having a sick baby

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-10-17 (Actual)

PRIMARY OUTCOMES:
Maternal sensitivity | Maternal sensitivity will be measured 3 months after the third NBO session at infant ages 4 months
  Maternal sensitivity is measured in the dyad of mother-infant communication; as appropriate responsiveness and ability to handle conflicts in the relationship. Scores for each subscale range from 1-7, higher scores indicating more sensitivity. Direct score range from 7-29, higher scores indicate more sensitivity. Direct score leads to Clinical-Screener score which is reated on a 100 point dimentional scale, divided into four zones; Emotional-Availability (81-100), Complicated E-A (61-80), Unavailable/Detached E-A (41-60) and Problematic/disturbed E-A (1-40).
  The EA Scale is validated in various settings and cultures and will serve as the main outcome measure in the RCT.
Childs responsiveness | Childs responsiveness will be measured 3 months after the third NBO session at infant ages 4 months
  Childs responsiveness is measured in the dyad of mother-infant communication; as willingness to respond to bids of the adult without over-compliance. Scores for each subscale range from 1-7, higher scores indicating more responsivenss. Direct score range from 7-29, higher scores indicate more responsiveness. Direct score leads to Clinical-Screener score which is rated on a 100 point dimentional scale, divided into four zones; Emotional-Availability (81-100), Complicated E-A (61-80), Unavailable/Detached E-A (41-60) and Problematic/disturbed E-A (1-40)

CONTACTS AND LOCATIONS:
Overall Officials: Anna M Jonsdottir, PhD, Study Director — team leader
Locations (1):
- Stefanía Birna Arnardóttir, Reykjavik, Ísland, Iceland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Valla L, Slinning K, Wentzel-Larsen T, Rosand GM, Arnardottir SB. The newborn behavioural observations (NBO) system embedded in routine postpartum care in at-risk families in Iceland: a randomised controlled trial. BMC Pregnancy Childbirth. 2025 Jan 8;25(1):13. doi: 10.1186/s12884-024-07128-0. PMID 39780054